CLINICAL TRIAL: NCT03020706
Title: Effect of Magnesium Sulphate on Neostigmine-induced Reversal of Neuromuscular Block by Rocuronium
Brief Title: Effect of Magnesium Sulphate on Neostigmine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Park Hee-Yeon, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: B-1610/367-002
Record Dates: First submitted 2017-01-08; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Neuromuscular Blockade
Keywords: magnesium sulphate; neostigmine
MeSH Terms: interventions — Magnesium Sulfate; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Experimental): magnesium sulfate, injectable intravenous administration (50mg/kg diluted in 100ml normal saline) during general anesthesia
  Interventions: Drug: Magnesium Sulfate, Injectable
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Magnesium Sulfate, Injectable — magnesium sulphate intravenous administration during general anesthesia
  Other Names: magnesium sulphate
  Arms: Magnesium

SUMMARY:
The purpose of this study is to evaluate the effect of magnesium sulphate on neostigmine-induced reversal of neuromuscular block by rocuronium

DETAILED DESCRIPTION:
Comparison of reversa time by neostigmine in magnesium group and control group

ELIGIBILITY:
Inclusion Criteria:

* ASA status 1 or 2
* patients undergoing surgery for more than 60 min under general anesthesia

Exclusion Criteria:

* electrolyte abnormalities
* medication on aminoglycoside, antiepileptic drug, magnesium
* underweight or obesity (BMI <18.5 or >30)
* renal insufficiency (Cr>1.4 mg/dl)
* AV block
* neuromuscular disease (ex: Myathenia gravis)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
reversal time | through study completion, an average of 90 minutes
  reversal time: from neostigmine injection to TOF ratio 0.9

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hwan Do, MD, Ph D, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Kyungi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided